CLINICAL TRIAL: NCT06424730
Title: Team Based Equity Conscious Telemedicine Approach to Improve Hypertension Among Black Patients
Brief Title: Team Based Equity Conscious Telemedicine Approach to Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: closed because we were funded for another similar study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00113617
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: high blood pressure; telemedicine; African-American
MeSH Terms: conditions — Hypertension | interventions — Methods; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study has two main objectives. First, to evaluate multi-level barriers and facilitators for recruitment and participation of Black patients in a TET-HTN clinical trial (Aim 1). Second objective is to evaluate the feasibility of TET-HTN intervention in a randomized comparison with usual clinic-based hypertension care approach (Aim 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interview Group (Other): Black patients or their family members; Black community faith leaders; primary care providers and research coordinators
  Interventions: Other: Feasibility Interview
- Team based Equity conscious Telemedicine Hypertension (TET-HTN) intervention (Experimental): Black patients with systolic blood pressure >140 mmHg on the last two clinic visits plus baseline systolic blood pressure >130 mmHg - deliver the TET-HTN intervention over six months
  Interventions: Behavioral: Team Based Equity Conscious Telemedicine Hypertension Intervention
- Usual Care (Other): Black patients with systolic blood pressure >140 mmHg on the last two clinic visits plus baseline systolic blood pressure >130 mmHg - usual clinic based hypertension care using routinely available clinic services including community health worker/social worker. Clinicians can offer self-management support (e.g., dietician referral) or recommend a home blood pressure monitor. These activities mirror current primary care practice.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Other: Feasibility Interview — One audio-recorded interview with the participants lasting about 30-minutes
  Other Names: One audio-recorded interview
  Arms: Interview Group
Behavioral: Team Based Equity Conscious Telemedicine Hypertension Intervention — Will provide blood pressure monitor connected to a telehealth application. Patients will be asked to measure home blood pressure once daily. Will intensify medications as needed based on blood pressure measurement. Trained nurses or pharmacists will provide 4 self-management telephone calls (up to 30 minutes per call) to patients to address hypertension knowledge, medication adherence, healthy eating, physical activity, weight management, stress management, tobacco and alcohol use, and sleep apnea (with referrals if needed). Will support needs relevant in blood pressure control using locally available resources via community health worker and social workers.
  Other Names: Team based Equity conscious Telemedicine Hypertension (TET-HTN) intervention
  Arms: Team based Equity conscious Telemedicine Hypertension (TET-HTN) intervention
Behavioral: Usual Care — Usual clinic based hypertension care using routinely available clinic services including community health worker/social worker. Clinicians can offer self-management support (e.g., dietician referral) or recommend a home blood pressure monitor. These activities mirror current primary care practice.
  Other Names: Standard of Care
  Arms: Usual Care

SUMMARY:
The purpose of study is to understand the different factors (patient, societal, provider, clinic, health system) relevant in recruitment and participation of patients in Team Based Equity Conscious Telemedicine Approach to Improve Hypertension clinical trial.

DETAILED DESCRIPTION:
Black patients suffer disproportionate hypertension (HTN) burden with worse control, resulting in HTN-related mortality rates twice those observed in non-Hispanic White patients. Contextually informed care approach is urgently needed in Black patients for HTN management. This study will evaluate multi-level barriers and facilitators for recruitment and participation of Black patients in a Team Based Equity Conscious Telemedicine Approach to Improve Hypertension (TET-HTN) clinical trial. This study will also evaluate the feasibility of TET-HTN intervention in a randomized comparison with usual clinic-based hypertension care approach.

ELIGIBILITY:
Inclusion Criteria:

* African American or Black
* Patients with last clinic systolic Blood Pressure >140 mmHg or diastolic Blood Pressure >90 mmHg or both

Exclusion Criteria:

* Unable to read or speak English
* diminished ability to measure home BP (dementia, or psychosis)
* acute health changes in past 3 months increasing chance of BP instability (hospitalization);
* terminal illness.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Barriers / Facilitators for Recruitment | Day 1
  Evaluate multi-level barriers and facilitators for recruitment and participation of Black patients in a Team based Equity conscious Telemedicine (TET-HTN) clinical trial - will be reported as themes from thematic analysis of qualitative data
Feasibility of Telemedicine Approach - Proportion of Subjects | Month 6
  Evaluate the feasibility of Team Based Equity Conscious Telemedicine Hypertension intervention in a randomized comparison with usual clinic-based hypertension care. Feasibility will be measured using the proportion of patients screened, eligible, agree to participate and decline.

SECONDARY OUTCOMES:
Change in Blood Pressure | Month 6
  Changes in Systolic and Diastolic Blood Pressure
Percentage of Medication adherence | Month 6
  Medication adherence using the Proportion of Days Covered

OTHER OUTCOMES:
Number of Emergency Department and Urgent Care Visits | Month 6
  Number of clinic, urgent care and emergency department visits
Number of Subjects using Blood Pressure Monitors | Month 6
  Patient self-reported home BP monitor use

CONTACTS AND LOCATIONS:
Overall Officials: Yashashwi Pokharel, MD, MSCR, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No